CLINICAL TRIAL: NCT00004317
Title: Phase IV Randomized Study of Pyrimethamine, Sulfadiazine, and Leucovorin Calcium for Congenital Toxoplasmosis
Brief Title: Pyrimethamine, Sulfadiazine, and Leucovorin in Treating Patients With Congenital Toxoplasmosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Chicago (Other)
Responsible Party: Rima McLeod, MD Professor, University of Chicago
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 199/11837; UCCRC-08796; MRH-850410; UCRCC-08796; NCT00170599 (obsolete NCT alias)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Toxoplasmosis
Keywords: immunologic disorders and infectious disorders; rare disease; toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Leucovorin; Pyrimethamine; Spiramycin; Sulfadiazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): This group of infants is treated with a loading dose of oral pyrimethamine followed by a higher dose for the first two months then a lower dose for the remainder of the 12 months. Sulfadiazine and leucovorin calcium are also given orally for 12 months. The pyrimethamine loading dose is omitted if prior prenatal therapy was given.
  Interventions: Drug: Leucovorin calcium; Drug: Pyrimethamine; Drug: Spiramycin; Drug: Sulfadiazine
- 2 (Experimental): This group of infants is treated with a higher dose of oral pyrimethamine for the first 6 months and then the lower dose for the remainder of the 12 months. Sulfadiazine and leucovorin calcium are administered concurrently.
  Interventions: Drug: Leucovorin calcium; Drug: Pyrimethamine; Drug: Spiramycin; Drug: Sulfadiazine

INTERVENTIONS:
Drug: Leucovorin calcium — See arm descriptions
Drug: Pyrimethamine — See arm descriptions
Drug: Spiramycin — Spiramycin is administered before the fetal diagnosis is made.
Drug: Sulfadiazine — See arm descriptions

SUMMARY:
RATIONALE: Congenital toxoplasmosis is an infection caused by the parasitic organism Toxoplasma gondii, and it may be passed from an infected mother to her unborn child. The mother may have mild symptoms or no symptoms; the fetus, however, may experience damage to the eyes, nervous system, skin, and ears. The newborn may have a low birth weight, enlarged liver and spleen, jaundice, anemia, petechiae, and eye damage. Giving the antiparasitic drugs pyrimethamine and sulfadiazine is standard treatment for congenital toxoplasmosis, but it is not yet known which regimen of pyrimethamine is most effective for the disease.

PURPOSE: Randomized phase IV trial to determine which regimen of pyrimethamine is most effective when combined with sulfadiazine and leucovorin in treating patients who have congenital toxoplasmosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Infants are randomly assigned to 1 of 2 treatment groups. Patients are stratified by disease severity, chorioretinitis, prenatal treatment, and certainty of diagnosis at birth.

One group of infants is treated with a loading dose of oral pyrimethamine followed by a higher dose for the first two months then a lower dose for the remainder of the 12 months. Sulfadiazine and leucovorin calcium are also given orally for 12 months. The pyrimethamine loading dose is omitted if prior prenatal therapy was given.

Another group of infants is treated with a higher dose of oral pyrimethamine for the first 6 months and then the lower dose for the remainder of the 12 months. Sulfadiazine and leucovorin calcium are administered concurrently.

Infected fetuses of pregnant women are nonrandomly assigned to treatment with pyrimethamine, sulfadiazine, and leucovorin calcium after the first trimester. Spiramycin is administered before the fetal diagnosis is made.

Concurrent prednisone for active retinal inflammation or elevated cerebrospinal fluid protein is allowed.

Collaborating physicians will also refer historical controls, who have not been treated in the first year of life or who received one month or less therapy, and are older than one year. Absence of treatment in the first year of life will be due to parental preference, prior inadequate follow-up by the family physicians, or lack of detection or treatment of eye disease before the age of one year in otherwise asymptomatic children. These historical, untreated patients (who enter the study when they are older than one year) will be compared with treated children in the randomized study. These historical patients will not be randomized. Any abnormality requiring treatment (e.g., active chorioretinitis) in any child (including historical patients) will be treated.

All infants are followed at birth, then at age 1, 3.5, 5, 7.5, 10, 15, and 20.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Infants with congenital toxoplasmosis Toxoplasma gondii confirmed prior to age 2.5 months
* Pregnant women with evidence of toxoplasma infection by clinical observation and amniotic fluid sampling
* Acute infection acquired during gestation with evidence of fetal infection
* Untreated older children entered as controls
* Asymptomatic congenital toxoplasmosis
* Age more than 1 year
* No treatment within the first year of life
* No more than 1 month of prior therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2000-07; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Persistent motor abnormality | At pre-specified time points
Vision | At pre-specified time points
Hearing | At pre-specified time points
New chorioretinal lesion | At pre-specified time points
IQ less than 70 | At pre-specified time points
Decrease in IQ of greater than or equal to 15 points | At pre-specified time points

CONTACTS AND LOCATIONS:
Overall Officials: Rima McLeod, Study Chair — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] McLeod R, Boyer KM, Lee D, Mui E, Wroblewski K, Karrison T, Noble AG, Withers S, Swisher CN, Heydemann PT, Sautter M, Babiarz J, Rabiah P, Meier P, Grigg ME; Toxoplasmosis Study Group. Prematurity and severity are associated with Toxoplasma gondii alleles (NCCCTS, 1981-2009). Clin Infect Dis. 2012 Jun;54(11):1595-605. doi: 10.1093/cid/cis258. Epub 2012 Apr 11. PMID 22499837